CLINICAL TRIAL: NCT02712021
Title: Effects of Lycra Suits in Children With Cerebral Palsy
Acronym: CP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catholic University, Italy (Other)
Responsible Party: Principal Investigator, Domenico Romeo, MD, PhD, Catholic University, Italy
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27711/14
Record Dates: First submitted 2016-03-09; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Lycra; Motor Function; Static Balance
MeSH Terms: conditions — Cerebral Palsy

ARMS (2):
- Cerebral Palsy-Study group (Experimental): The intervention consisted of wearing a lycra suit, with shoulder, trunk and pelvis coverage, for more than 4 hours per day for 6 months. The motor function assessments will be performed without the Lycra suit, whereas the static balance assessments were performed with and without the suit.
  Interventions: Other: Lycra suit and physiotherapy treatment
- Cerebral Palsy-Control Group (Active Comparator): Children with clinical characteristics similar to the study group; they will be assessed using the same protocol but with no use of lycra garments
  Interventions: Other: physiotherapy treatment

INTERVENTIONS:
Other: Lycra suit and physiotherapy treatment — Garments will be fitted by an occupational therapy with the treating therapist and child neurologist present. The garments will be constructed of Lycra with the possibility of adding reinforcing panels or derotation bands. All the children will be involved in regular physiotherapy treatment (2-3/week).
  Arms: Cerebral Palsy-Study group
Other: physiotherapy treatment — All the children will be involved in regular physiotherapy treatment (2-3/week).
  Arms: Cerebral Palsy-Control Group

SUMMARY:
Lycra garments have recently been used for children with cerebral palsy, with favorable effects on alignment, biomechanics and neuromuscular activity. The aim of the present study is to determine the efficacy of a Lycra suit in improving motor function and static balance in children with cerebral palsy. The children included in this study will be part of a prospective project on children with cerebral palsy, older than 4 years of age, and their families regularly followed at the Child Neurology Unit of the Catholic University of Rome.

DETAILED DESCRIPTION:
A total of 10 children with cerebral palsy will be recruited and included in the study. Five of them will be considered as study group and will wear a lycra suit, with shoulder, trunk and pelvis coverage, for more than 4 hours per day for 6 months. The other 5 will be considered as control group, matched for age and sex to the study group, and will not wear the lycra suit. The evaluation of static balance and the gross motor function measure will be used as outcome measure. The children of both groups will be assessed twice, at baseline and 6 months after, each child acting as his/her own control.

The motor function assessments will be performed without the Lycra suit, whereas the static balance assessments were performed with and without the suit.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cerebral palsy based on the predominant type of motor impairment and classified according to the criteria proposed by Himmelmann.

Exclusion Criteria:

* Presence of major congenital malformations or metabolic or haematological complications.
* The investigators will also exclude children who had previously worn a lycra garment and who received Botulinum toxin injections or orthopaedic surgery in the year before the study.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline evaluation of static balance at 6 months | The children were assessed twice, at baseline and 6 months after, each child acting as his/her own control.
  The evaluation of static balance will be assessed by a "seated stabilometry exam" performed on a "Prokin PK 254 P" device produced by TecnoBody S.r.l. (Dalmine BG - Italy). This device consists of a static plate (47 centimeters of circumference) equipped internally with four piezoelectric sensors positioned at the extremity of the four cardinals points.

SECONDARY OUTCOMES:
Change from baseline Gross Motor Function Classification System at 6 months | The children were assessed twice, at baseline and 6 months after, each child acting as his/her own control.
  The Gross Motor Function Measure (GMFM) will be used to evaluate gross motor function quantitatively. The GMFM consists of 88 items grouped into 5 dimensions: A (lying and rolling), B (sitting), C (crawling and kneeling), D (standing), E (walking, running and jumping). Scores for each dimension are expressed as a percentage of the maximum score for that dimension. A total score is obtained by adding the scores for all dimensions and dividing by 5, ranging from 0 to 100.

REFERENCES:
- [Result] Himmelmann K, Hagberg G, Beckung E, Hagberg B, Uvebrant P. The changing panorama of cerebral palsy in Sweden. IX. Prevalence and origin in the birth-year period 1995-1998. Acta Paediatr. 2005 Mar;94(3):287-94. doi: 10.1111/j.1651-2227.2005.tb03071.x. PMID 16028646
- [Result] Flanagan A, Krzak J, Peer M, Johnson P, Urban M. Evaluation of short-term intensive orthotic garment use in children who have cerebral palsy. Pediatr Phys Ther. 2009 Summer;21(2):201-4. doi: 10.1097/PEP.0b013e3181a347ab. PMID 19440130
- [Result] Matthews MJ, Watson M, Richardson B. Effects of dynamic elastomeric fabric orthoses on children with cerebral palsy. Prosthet Orthot Int. 2009 Dec;33(4):339-47. doi: 10.3109/03093640903150287. PMID 19961295